CLINICAL TRIAL: NCT03003013
Title: Effect of Biphasic Bone Graft Material (BGM) in Combination With Autologous Platelet-rich Fibrin (PRF) on Bone Regeneration in an Odontogenic Maxillary Cyst: a Randomized Clinical Trial
Brief Title: Effect of Biphasic Bone Graft Material With Autologous Platelet-rich Fibrin on Bone Regeneration in a Maxillary Cyst
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherif Abdel Monem Abdel Aziz, Master student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CU
Record Dates: First submitted 2016-11-16; First posted 2016-12-26 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Odontogenic Maxillary Cysts
Keywords: Odontogenic cysts; Bone substitutes materials; SYMBIOS®; Platelets rich fibrin (PRF); Bone regeneration
MeSH Terms: conditions — Odontogenic Cysts

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biphasic Bone Graft With Autologous Platelet-rich Fibrin (Active Comparator): Patients will undergo complete removal of the cystic cavity with the application of SYMBIOS biphasic bone graft material in combination with PRF in the cystic cavity
  Interventions: Procedure: Biphasic Bone Graft Material (BGM) in Combination With Autologous Platelet-rich Fibrin (PRF)
- Biphasic Bone Graft Material only (Active Comparator): Patients will undergo complete removal of the cystic cavity with the application of SYMBIOS biphasic bone graft material without PRF in the cystic cavity
  Interventions: Procedure: Biphasic Bone Graft Material (BGM) in Combination With Autologous Platelet-rich Fibrin (PRF)

INTERVENTIONS:
Procedure: Biphasic Bone Graft Material (BGM) in Combination With Autologous Platelet-rich Fibrin (PRF)

SUMMARY:
Effect of Biphasic Bone Graft Material (BGM) in combination with autologous platelet-rich fibrin (PRF) on bone regeneration in an odontogenic maxillary cyst: a randomized clinical trial

DETAILED DESCRIPTION:
Odontogenic cysts are the most common form of cystic lesions that affect the oral and maxillofacial region. Their origin, mechanism of growth, as well as treatment problems have been often discussed.

Platelet rich fibrin (PRF) is a second generation platelet concentrate first developed in France by Choukron et al in 2001, prepared from centrifuged autologous blood. It is a fibrin clot rich in platelets without addition of bovine thrombin, calcium chloride or anticoagulant during preparation thus eliminating the risks associated with the use of thrombin. Platelet rich fibrin is derived from a natural and progressive polymerization occurring centrifugation. A progressive or relatively slow polymerization mode may increase incorporation of the circulating cytokines in the fibrin meshes which are then released in a relatively long-term and controllable way which in turn will help in soft tissue healing and accelerated bone regeneration.

Blood Derivatives Enhancing Bone Regeneration:

1-Fibrin glue: It is classically described as a two component mixture in which concentrated fibrinogen factor XIII and fibronectin are added to thrombin ,calcium choloride and an inhibitor of fibrinolysis to form a fibrin clot .

Shortcomings:

The risk of transmission of virus, like human immunodeficiency virus (HIV). 2. Autologous Fibrin Adhesives: The patient's blood is harvested 1:3 weeks before the intervention and requires separating one unit of whole blood cell component and plasma fraction for use as cryoprecipitate.

Shortcomings:

* Extremely long.
* Complex protocols. 3. Platelet rich plasma (PRP): It is a modification type of autologous fibrin adhesives which requires autologous blood collection in the immediate preoperative period and processing in the centrifugation which is then mixed with bovine thrombine and calcium chloride at the time of application.

Shortcomings:

1. The use of bovine thrombin puts the patient at risk of life -threating coagulopathies associated with the development of antibodies to factor V , XI and thrombin .
2. Higher concentration of thrombin impedes cell migration during bone healing.
3. It mediates only the early aspects of bone repair. A variety of treatment modalities including the use of autogenous bone grafts and bone substitutes materials ,guided tissue regeneration (GTR) with the use of barrier membranes and growth factors have been used to stimulate bone regeneration mechanism.The drawbacks associated with autogenous bone grafts have led to the production of a large number of alternative bone substitute materials. Their biological behavior depends upon their chemical composition and physicochemical structure. Bone grafting materials include autografts, allografts, xenografts and alloplasts. The osteoconductive hydroxyapatite grafting materials have been widely used to enhance new bone regeneration.

SYMBIOS®:

Biphasic Bone Graft Material (BGM) is a resorbable inorganic bone forming material in granular form of plant origin derived from red marine algae. The chemical composition of this interconnected porous biological product is similar to the inorganic part of the human bone. It is a composition of 20% hydroxyapatite (HA) and 80% β-tricalciumphosphate (ß-TCP). Due to the high tricalcium- phosphate content of the product it resorbs significantly faster than pure hydroxyapatite. The biphasic BGM is biocompatible and osteoconductive. The selection of the two grain sizes is dependent on the defect.

Growth factors represent an area of interest for surgeons attempting to modify and enhance the wound healing process and tissue regeneration. However, the Platelet-Rich Plasma (PRP) is already in use for some time by hematologists for transfusions and prevention of bleeding episodes in patients with severe thrombocytopenia.

Uses of PRF Over PRP:

1. The improved mechanical properties of PRF over conventional PRP translate it into a biologic matrix that is easy to handle and implant in awide variety of tissue repair applications.
2. Platelets rich fibrin has increased modulus of elasticity. This property imparts it better pliability and drapability, allowing it to closely conform to awide variety of irregular surgical sites and surfaces similar to split thickness skin auto grafts.
3. Platelet rich fibrin can easily be sutured to surgical site.

Benefits of this study to patients:

* Treatment of cystic lesions.
* Enhancement of bone regeneration.

Benefits of this study for other clinicians:

The study provides a new modality for the regeneration of new bone after cystic enucleation.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria

1. Age range is 15: 60 years old.
2. A maxillary odontogenic cysts larger than 3 cm in size.

Exclusion criteria

1. A maxillary odontogenic cysts smaller than 3 cm in size.
2. A mandibular odontogenic cysts.
3. Non odontogenic cysts.
4. Patients with thrombotic risk factors or taking anti-platelets drugs.
5. Patients with systemic diseases

Exclusion Criteria:

-

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Swelling | six weeks
  Visual analogue scale

SECONDARY OUTCOMES:
bone regeneration | from six to nine months
  Gray scale value via cone beam CT

CONTACTS AND LOCATIONS:
Overall Officials: Niven Abal Latif Askar, PhD, Study Director — Assistant Professor of Oral& Maxillofacial Surgery
Locations (1):
- Faculty of Oral & Dental Medicine Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No